CLINICAL TRIAL: NCT01018420
Title: A Randomized, Double-Blind, Double-Dummy Pharmacokinetic and Exploratory Electrocardiogram (ECG) Safety Study of a Standard Acute Gout Regimen
Brief Title: Pharmacokinetic and Exploratory Electrocardiogram (ECG) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MPC-004-07-1002
Record Dates: First submitted 2009-08-12; First posted 2009-11-23 (Estimated); Results first posted 2009-11-23 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Pharmacokinetics
Keywords: healthy
MeSH Terms: interventions — Colchicine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colchicine (Experimental)
  Interventions: Drug: Colchicine
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Colchicine — two 0.6 mg capsules (1.2 mg dose) followed by an additional 0.6mg capsule every hour for 6 additional doses
  Other Names: COLCRYS TM
  Arms: Colchicine
Drug: Moxifloxacin — 400 mg capsule at the 6 hour point
  Arms: Moxifloxacin

SUMMARY:
This study will characterize the pharmacokinetics of colchicine after an oral dosing regimen of 4.8 mg over 6 hours. In addition it will compare the electrocardiogram (ECG) changes, if any, from this dosing regimen to that of a single dose of moxifloxacin 400 mg, a positive control for the corrected QT interval (QTc) prolongation.

DETAILED DESCRIPTION:
This study will characterize the pharmacokinetics of colchicine after an oral dosing regimen of 4.8 mg over 6 hours. In addition, it will determine whether or not there is a trend toward effect of this high dose regimen on the electrocardiogram (ECG), mainly the corrected QT interval (QTc), via comparison to a 400 mg dose of moxifloxacin, a positive control for QTc prolongation. Eighteen healthy, non-smoking, non-obese, non-pregnant adults between the ages of 18 to 55 years of age will be randomized in a double blind fashion to either the colchicine or moxifloxacin treatment groups. On the day prior to the study (Day -1), subjects will receive colchicine and moxifloxacin placebos according to the same schedule and conditions as will be present during the study, and baseline ECG's will be determined by 24 hour 12-lead Holter monitoring. On Day 1, after a minimum 10 hour overnight fast, subjects enrolled in the colchicine treatment group (N=15) will receive two 0.6 mg capsules (plus one dose moxifloxacin placebo) followed by an additional 0.6 mg colchicine dose (plus one dose moxifloxacin placebo) every hour for 6 additional doses; subjects in the moxifloxacin treatment group will receive placebo doses matching the colchicine treatment group over the first 5 hours, then 400 mg moxifloxacin (plus one dose colchicine placebo) at the 6 hour point. Fasting will continue for 4 hours after the first dose at which time a standardized meal will be served. Blood will be drawn from all participants at times sufficient to adequately define the pharmacokinetics of colchicine. During the study, continuous 24-hour ECG monitoring via 12-lead Holter monitor will be performed. Triplicate ECG records will be extracted from 5 minute observation periods throughout the 24 hours post dose. Finally, all study subjects will be monitored for adverse effects throughout the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-55 years of age, non smoking and non-pregnant, weighing at least 55kg and within 15% of ideal body weight, with no significant EKG changes

Exclusion Criteria:

* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease
* History or family history of congenital long QT syndrome (LQTS) or sudden death possibly related to LQTS
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 30 days prior to the first dose and throughout the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, Pharm.D., Principal Investigator — PRACS Institiute, Ltd.
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighteen (18) healthy, non-smoking, adult male and female volunteers, consisting of university students and members of the community at large, were to be enrolled.
Pre-assignment Details: 50 subjects screened, 28 were screen failures, 4 were alternates
Groups:
- Colchicine: 1.2mg initially (two 0.6 mg capsules) followed by an additional 0.6mg capsule every hour for 6 additional doses [4.8mg over 6 hours]
Period: Overall Study
Arm/Group | Colchicine | Moxifloxacin
Started | 15 | 3
Completed | 15 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colchicine | Moxifloxacin | Total
Number analyzed (Participants) | 15 | 3 | 18
Age, Categorical [Count of Participants; unit: Participants] — age range: >=18 and <=55
  Participants
    <=18 years | 0 | 0 | 0.0
    Between 18 and 65 years | 15 | 3 | 18.0
    >=65 years | 0 | 0 | 0.0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.1 (10.4) | 21.3 (0.6) | 28.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8.0
  Male | 8 | 2 | 10.0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1.0
  Asian | 0 | 0 | 0.0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0.0
  Black or African American | 1 | 0 | 1.0
  White | 13 | 3 | 16.0
  More than one race | 0 | 0 | 0.0
  Unknown or Not Reported | 0 | 0 | 0.0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 3 | 18.0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that colchicine reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples collected pre-dose and 1 (prior to second dose), 3 (prior to fourth dose), 6 (prior to final dose), 6.17, 6.33, 6.5, 6.75, 7, 7.25, 7.5, 7.75, 8, 10, 12, 23, 36, 48, 72 and 96 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Colchicine
Number analyzed (Participants) | 15
ng/mL | 6.84 (1.30)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Colchicine
Number analyzed (Participants) | 15
ng-hr/mL | 104.95 (24.61)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Colchicine
Number analyzed (Participants) | 15
ng-hr/mL | 118.20 (26.01)

4. Secondary Outcome: Electrocardiogram (ECG) Evaluation of the QTcF Interval (Colchicine)
Description: The QT interval assesses cardiac repolarization and risk for arrhythmias. It is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. It is dependent on heart rate and is corrected (c) to aid interpretation via Fridericia's adjustment (F), and is reported as QTcF.
Time Frame: 24 hours - measured 0.5 hr prior to first dose (baseline), then 1, 3, 6, 7, 8, 10, 12, and 23 hours after first dose
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Baseline: measured 0.5 hr prior to initial colchicine dose
- Hour 1: measured 1 hour after initial colchicine dose
- Hour 3: measured 3 hours after initial colchicine dose
- Hour 6: measured 6 hours after initial colchicine dose
- Hour 7: measured 7 hours after initial colchicine dose
- Hour 8: measured 8 hours after initial colchicine dose
- Hour 10: measured 10 hours after initial colchicine dose
- Hour 12: measured 12 hours after initial colchicine dose
- Hour 23: measured 23 hours after initial colchicine dose
Arm/Group | Baseline | Hour 1 | Hour 3 | Hour 6 | Hour 7 | Hour 8 | Hour 10 | Hour 12 | Hour 23
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15
milliseconds | 401.62 (20.18) | 397.80 (19.63) | 401.76 (20.04) | 394.73 (10.72) | 388.84 (15.57) | 393.93 (16.30) | 396.02 (16.15) | 396.89 (11.85) | 399.36 (17.38)

5. Secondary Outcome: Electrocardiogram (ECG) Evaluation of the QTcF Interval (Moxifloxacin)
Description: as for outcome 4
Time Frame: 24 hours - measured 0.5 hr prior to dose (baseline), then 1, 3, 6, 7, 8, 10, 12, and 23 hours after dose
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Baseline: measured 0.5 hour prior to moxifloxacin dose
- Hour 1: measured 1 hour after moxifloxacin dose
- Hour 3: measured 3 hours after moxifloxacin dose
- Hour 6: measured 6 hours after moxifloxacin dose
- Hour 7: measured 7 hours after moxifloxacin dose
- Hour 8: measured 8 hours after moxifloxacin dose
- Hour 10: measured 10 hours after moxifloxacin dose
- Hour 12: measured 12 hours after moxifloxacin dose
- Hour 23: measured 23 hours after moxifloxacin dose
Arm/Group | Baseline | Hour 1 | Hour 3 | Hour 6 | Hour 7 | Hour 8 | Hour 10 | Hour 12 | Hour 23
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
milliseconds | 402.11 (12.04) | 398.89 (1.65) | 403.67 (17.91) | 397.00 (8.46) | 397.89 (8.31) | 397.44 (2.59) | 402.67 (13.23) | 405.22 (17.64) | 416.00 (13.68)

ADVERSE EVENTS:
Arm/Group | Colchicine | Moxifloxacin
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/3
Other Adverse Events (participants affected / at risk) | 15/15 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine (N=15) | Moxifloxacin (N=3)
diarrhoea (Gastrointestinal disorders) | 15 (15) | 0 (0)
flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 7 (7) | 0 (0)
vessel puncture site pain (General disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 6 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days